CLINICAL TRIAL: NCT01016210
Title: The Effect of Luteinizing Hormone (LH) Supplementation Following Gonadotropin-releasing Hormone (GnRH) Antagonist Administration in Advanced Reproductive Ageing Women Undergoing IVF and Embryo Transfer (IVF/ET)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Baruch Padeh Medical Center, Poriya (Other Government)
Collaborators: Ministry of Health, Israel (Other Government)
Responsible Party: DR Joni Younis, The baruch Padeh Medical center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Leuveris1.CTIL
Record Dates: First submitted 2009-11-18; First posted 2009-11-19 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2014-01

CONDITIONS: Pregnancy Result Rape
Keywords: pregnancy; IVF

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 60 infertile women (Experimental): Candidates for IVF-ET treatment
  Interventions: Drug: Leuveris
- control (No Intervention): no treatment

INTERVENTIONS:
Drug: Leuveris — IV
  Arms: 60 infertile women
Drug: Leuveris — All recruited women will be treated similarly employing the recombinant FSH and the fixed GnRH antagonist. Concomitantly, on the same day of the antagonist administration r-LH will be administered daily and continued until human chorionic gonadotropin (hCG) day.
  Arms: 60 infertile women

SUMMARY:
To explore whether recombinant LH (rLH) supplementation (Leuveris) to recombinant follicle stimulating hormone (rFSH) following GnRH antagonist treatment has an advantage in infertile women with advanced reproductive ageing undergoing IVF-ET.

ELIGIBILITY:
Inclusion Criteria:

* female candidate to IVF
* between 30-45 years old

Exclusion Criteria:

* not included for fertilization

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-02; Primary Completion 2012-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Pregnancy rate | Starting February 2010

SECONDARY OUTCOMES:
Fertilization rate | Starting February 2010 till April 2013

CONTACTS AND LOCATIONS:
Locations (1):
- Poriya hospital, Tiberias, Israel